CLINICAL TRIAL: NCT00733122
Title: Evaluation of Tolerability and Immunogenicity of GARDASIL in Healthy Females, Between 16 and 26 Years of Age, in India.
Brief Title: Tolerability and Immunogenicity of Gardasil in Females Between 16 and 23 Years of Age in India (V501-034)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Following the direction of the local (India) health authority, data specified in the protocol were not collected and study was cancelled.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V501-034; 2008_016 (Other: Merck Registration Number); CTRI/2009/091/000787 (Registry Identifier: CTRI)
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: HPV Infections
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

ARMS (1):
- A (Experimental): GARDASIL, Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine
  Interventions: Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine

INTERVENTIONS:
Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine — Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine 0.5 mL of GARDASIL as intramuscular injections at the Day 1, Month 2, and Month 6 visits.

SUMMARY:
This study is designed to determine the tolerability and immunogenicity of a 3-dose regimen of Gardasil administered to healthy married females between 16 and 23 years of age, in India.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Married Females Between 16 And 23 Years Of Age With Intact Uteri
* No Clinical Evidence Of Gross Purulent Cervicitis (Otherwise Postpone Until After Treatment Or Lack Of Laboratory Confirmation Of Treatable Cause
* Must Agree To Refrain From Sexual Activity (Including Vaginal And Anal Penetration And Any Genital Contact) For 48 Hours Prior To Any Scheduled Visit That Includes A Pelvic Examination In An Attempt To Avoid Detection Of Viral DNA Which Has Been Deposited In The Vagina Or On The Perineal/Perianal Area During Sexual Intercourse And Is Not The Result Of Ongoing Infection
* Not Pregnant Now (As Determined By A Serum Pregnancy Test Or Urine Pregnancy Test Sensitive To 25 IU/L hCG), And Must Agree To Use Effective Contraception Through Month 7 Of The Study
* Must Agree To Provide Study Personnel With A Primary Telephone Number As Well As An Alternate Telephone Number For Follow-Up Purposes.
* Individuals Who Have Had Sexual Intercourse In The 2 Weeks Prior To Enrollment Must Have Been Using Effective Contraception As Defined Above (Emergency Contraception Is Not Considered Effective Contraception For Enrollment Into The Study.)

Exclusion Criteria:

* Individuals Concurrently Enrolled In Clinical Studies Of Investigational Agents Or Studies Involving Collection Of Cervical/Genital Specimens
* Feverish Feeling Within 24 Hours Prior To The First Injection And No Temperature < 100°F Or < 37.8°C (Oral Or Oral Equivalent) At First Vaccination
* History Of Recent Or Ongoing Alcohol Or Other Drug Abuse. Alcohol Abusers Are Defined As Those Who Drink Despite Recurrent Social, Interpersonal, And Legal Problems As A Result Of Alcohol Use
* History Of Known Prior Vaccination With An Hpv Vaccine Subject Has Received Non-Replicating (Inactivated) Vaccine Within 14 Days Prior To The Day 1 Vaccination Or Has Received Replicating (Live Virus) Vaccine Within 21 Days Prior To The Day 1 Vaccination
* Individuals With Any Prior Abnormal Pap Test Showing Squamous Intraepithelial Lesion (Sil), Ascus, Asc-Us, Asc-H Individuals With A History Of Genital Warts
* Individuals Allergic To Any Vaccine Component, Including Aluminium, Yeast, Or Benzonase™ (Nuclease, Nycomed [Used To Remove Residual Nucleic Acids From This And Other Vaccines])
* Individuals Who Have Received Any Immune Globulin Preparation Or Blood-Derived Products Within The 3 Months Prior To The First Injection, Or Plan To Receive Any Through The Completion Of The Study
* Individuals With A History Of Splenectomy, Known Immune Disorders (E.G., Systemic Lupus Erythematosus, Rheumatoid Arthritis), Or Receiving Immunosuppressives (E.G., Substances Or Treatments Known To Diminish Immune Response Such As Radiation Therapy, Administration Of Antimetabolites, Antilymphocytic Sera, Systemic Corticosteroids)
* Individuals Who Have Received Periodic Treatments With Immunosuppressives, Defined As At Least 3 Courses Of Systemic Corticosteroids Each Lasting At Least 1 Week In Duration For The Year Prior To Enrollment, Will Be Excluded. Subjects Using Topical Steroids (I.E., Inhaled Or Nasal) Will Be Eligible For Vaccination
* Individuals Who Are Immunocompromised Or Have Been Diagnosed As Having HIV Infection
* Individuals With Known Thrombocytopenia Or Any Coagulation Disorder That Would Contraindicate Intramuscular Injections
* Any Condition Which In The Opinion Of The Investigator Might Interfere With The Evaluation Of The Study Objectives
* Any Plans To Permanently Relocate From The Area Prior To The Completion Of The Study Or To Leave For An Extended Period Of Time When Study Visits Would Need To Be Scheduled
* Inability To Give Consent/Assent

Ages: 16 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2013-10-01 (Estimated); Study Completion 2013-10-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects who seroconvert to each of HPV 6, 11, 16, 18 at Week 4 Post dose 3 (Month 7), Month 24 and Month 36. | Week 4 Post dose 3 (Month 7), Month 24 and Month 36

SECONDARY OUTCOMES:
The Geometric Mean Titers (GMTs) | Week 4 Post dose 3 (Month 7), Month 24 and Month 36

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC